CLINICAL TRIAL: NCT05415358
Title: A Prospective Study Of Immune Signatures In Metastatic Non-Small Cell Lung Cancer (mNSCLC) Patients At Completion Of Immune Checkpoint Inhibitor Treatment Either As Monotherapy Or In Combination With Chemotherapy In The First Line Setting
Brief Title: Immune Signature Analysis of Disease Progression in Post Immunotherapy Lung Cancer Patients
Status: Active, not recruiting | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Atrium Health Levine Cancer Institute (Other); Atrium Health Wake Forest Baptist (Other)
Responsible Party: Sponsor
Other Study IDs: LCI-LUN-IMM-BIO-001; Pro00058707 (Other: Advarra IRB)
Record Dates: First submitted 2021-12-06; First posted 2022-06-13 (Actual); Last update posted 2026-02-03 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer, Nonsmall Cell
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Subjects will be given the option to consent to have any additional blood specimens retained for future unplanned research.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single Arm: Biomarkers and ctDNA data generated from patients with metastatic non-small cell lung carcinoma who have completed first line immune checkpoint inhibitor monotherapy or immune checkpoint inhibitor platinum doublet combination therapy, and have, at immunotherapy discontinuation, completed at least 20 of an anticipated 24 months of immune checkpoint inhibitor treatment.
  Interventions: Other: Blood and tissue samples

INTERVENTIONS:
Other: Blood and tissue samples — Blood and tissue will be collected to perform ctDNA and immune biomarkers assessment to predict progression within 6 months of immune checkpoint inhibitor treatment discontinuation.

SUMMARY:
The purpose of this study is to examine the association between ctDNA/immune biomarkers and disease progression in patients who, at immunotherapy discontinuation, have completed at least 20 of an anticipated 24 months of immune checkpoint inhibitor monotherapy or immune checkpoint inhibitor combination chemotherapy for mNSCLC.

DETAILED DESCRIPTION:
This is a prospective, non-randomized, pilot study. The target population is adults ≥18 years of age with metastatic non-small cell lung cancer that at immunotherapy discontinuation, have completed at least 20 of an anticipated 24 months of planned doses of immune checkpoint inhibitor treatment in the first line setting. The study will be conducted at various Atrium Health Wake Forest Baptist Comprehensive Cancer Center locations. Subjects will have blood for ctDNA and immune markers collected at baseline, and every 3 months for up to approximately 6 months. Blood will be collected at disease progression if it occurs prior to 6 months, ensuring that the collection occurs prior to start of subsequent anti-cancer therapy. We will also collect data from standard of care CT scans every 3 months for up to 6 months or until disease progression. In patients undergoing standard of care biopsies, a portion of tumor tissue will be obtained and tested for tumor mutations. Archived tumor tissue collected pre-immunotherapy (if available) will also be tested.

ELIGIBILITY:
Inclusion Criteria

1. Informed consent and HIPAA authorization for release of personal health information signed by the subject. Note: Data from tumor samples, blood samples and radiographic scans prior to enrollment date may be used.
2. Age greater than or equal to18 years at the time of consent.
3. Patients with metastatic non-small cell lung carcinoma have completed first line who, at immunotherapy discontinuation, have completed at least 20 of an anticipated 24 months of immune checkpoint inhibitor monotherapy or pembrolizumab combination chemotherapy in the first line setting.
4. Patients are allowed to continue maintenance chemotherapy.
5. Ability to understand and comply with study procedures for the entire length of the study.
6. Known PD-L1 prior to initiation of first-line treatment for NSCLC.

Exclusion Criteria

1. Enrollment/collection of baseline sample earlier than 7 days prior to scheduled last dose of immune checkpoint inhibitor treatment or more than 30 days after last dose of immune checkpoint inhibitor treatment.
2. Patients whose tumors harbor known first line treatment druggable gene abnormalities (e.g. EGFR, BRAF, ALK, ROS1).
3. Patients who have ever received or are currently receiving other types of immunotherapies (nivolumab, ipilimumab, durvalumab or atezolizumab).
4. Known pregnancy.
5. Patients who progress per the enrolling investigator while on treatment with immune checkpoint inhibitor treatment prior to enrollment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic non-small cell lung carcinoma who have completed first line immune checkpoint inhibitor monotherapy or immune checkpoint inhibitor platinum doublet combination therapy, and have, at immunotherapy discontinuation, completed at least 20 of an anticipated 24 months of immune checkpoint inhibitor treatment. These treatments are managed according to standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 23 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2035-09 (Estimated); Study Completion 2035-09 (Estimated)

PRIMARY OUTCOMES:
Disease progression status for the purpose of assessing its correlation with ctDNA measured at 0 months after pembrolizumab treatment completion | 6 months after immune checkpoint inhibitor treatment completion
  Disease progression status determined by the treating investigator per standard care

SECONDARY OUTCOMES:
Disease progression status for the purpose of assessing its correlation with circulating effector T cell anergy at 0 months after pembrolizumab treatment completion | 6 months after immune checkpoint inhibitor treatment completion
  Disease progression status determined by the treating investigator per standard care
Disease progression status for the purpose of assessing its correlation with the rate of effector to central memory T cell conversion at 0 months after pembrolizumab treatment completion | 6 months after immune checkpoint inhibitor treatment completion
  Disease progression status determined by the treating investigator per standard care
Disease progression status for the purpose of assessing its correlation with clonal circulating T cell diversity at 0 months after pembrolizumab treatment completion | 6 months after immune checkpoint inhibitor treatment completion
  Disease progression status determined by the treating investigator per standard care

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Mileham, MD, Principal Investigator — Atrium Health Levine Cancer
Locations (2):
- United States (2):
  - Atrium Health Levine Cancer, Charlotte, North Carolina
  - Atrium Health Wake Forest Baptist Comprehensive Cancer Center, Winston-Salem, North Carolina